CLINICAL TRIAL: NCT02436343
Title: Cardiac Performance in Pregnant Obese Women:Are They in Jeopardy?
Status: Completed | Type: Observational
Sponsor: Benha University (Other)
Collaborators: Armed Forces Hospitals, Southern Region, Saudi Arabia (Other Government)
Responsible Party: Principal Investigator, ahmed abdulmoneim altraigey, lecturer, Benha University
Other Study IDs: AFHSRMREC/2015/OB/GYNAE/061
Record Dates: First submitted 2015-05-02; First posted 2015-05-06 (Estimated); Last update posted 2018-07-11 (Actual); Status verified 2018-07

CONDITIONS: Cardiac Performance
Keywords: left ventricular functions; pregnancy; obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- obese pregnant women: pregnant women wit body mass index more than or equal to 30 kg/m2 will be subjected to four serial echocardiograms in the 3 trimesters of pregnancy and in the postpartum state.
  Height, weight, systolic and diastolic blood pressures will be measured at each echocardiographic evaluation.
  Interventions: Other: echocardiogram
- lean pregnant women: pregnant women wit body mass index less than or equal to 25kg/m2 will be subjected to four serial echocardiograms in the 3 trimesters of pregnancy and in the postpartum state.
  Height, weight, systolic and diastolic blood pressures will be measured at each echocardiographic evaluation.
  Interventions: Other: echocardiogram

INTERVENTIONS:
Other: echocardiogram — At each echocardiographic evaluation, the investigator will obtain the following parameters:
  Left ventricular internal dimensions at end diastole Left ventricular posterior wall thickness Left ventricular end systolic stress Left ventricular fractional shortening Velocity of circumferential shortening Left ventricular mass Contractility and indices of preload Stroke volume

SUMMARY:
The aim of this work is to Assess serial changes in "cardiovascular function" in morbidly obese pregnant females (BMI equal or higher than 30 kg/m2) as compared to normal lean pregnant female controls.

DETAILED DESCRIPTION:
Overweight and obesity are defined as: abnormal or, excessive fat accumulation that presents a risk to health. A crude population measure of obesity is the body mass index (BMI), a person's weight (in kilograms) divided by the square of his or her height (in meters). A person with a BMI of 30 or more is generally considered obese. A person with a BMI equal to or more than 25 is considered overweight.

Obesity has reached particularly alarming levels in the Middle East and North Africa (MENA) region. The prevalence of female obesity currently estimated at over 40% , had already exceeded that in Europe and the USA.

Obesity has been linked to several major chronic diseases, including type II diabetes, cardiovascular diseases, selected cancers, gallbladder disease, asthma, osteoarthritis, and chronic back pain.

Obesity has been also linked to a wide spectrum of cardiovascular changes ranging from a hyper dynamic circulation, through subclinical cardiac structural changes, to overt heart failure.

Obesity is associated with hemodynamic overload due to the increased metabolic demand imposed by the expanded adipose tissue and augmented fat-free mass in obesity results in a hyper dynamic circulation with increased blood volume. In addition to the increased preload, left ventricular (LV) after load is also elevated in obese individuals due to both increased peripheral resistance and greater conduit artery stiffness. Right ventricular after load may be increased, presumably due to associated sleep disordered breathing and LV changes.

Pregnancy is associated with hemodynamic and hormonal changes that can affect the heart. From the first trimester, there is an increase in cardiac output that places a volume load on the heart. Hormonal changes include increased circulating estrogen and relaxin, which may directly or indirectly affect the heart. During pregnancy, the heart undergoes remodeling similar to that observed in athletes, with increases in chamber dimensions, left ventricular (LV) wall thickness, and mass, that is consistent with a process of eccentric hypertrophy.

Myocardial contractile function also changes in pregnancy. Ejection-phase indices of LV function, including systolic fractional shortening (FS) and mean velocity of circumferential fiber thickening (V CFC), have been variously reported to increase, remain constant,or decrease, during pregnancy. Thus, obese women are more likely to encounter problems on becoming pregnant.

There is large evidence in the literature demonstrating that women who are overweight are at greater risk of developing pregnancy complications and problems associated with labor and delivery.

ELIGIBILITY:
Inclusion Criteria:

* Any pregnant woman in her 1st trimester with a singleton live healthy pregnancy

Exclusion Criteria:

* Multiple gestations.
* Anemia.
* Medical history of hypertension.
* Medical history of any cardiac disease.
* Medical history of pre-gestational diabetes.
* Development of gestational diabetes and pre-eclampsia.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Any pregnant woman in her 1st trimester with a singleton live healthy pregnancy will be eligible for inclusion in the study. Eligible women will be further categorized into case and control groups. Women with body mass index equals or more than 30kg/m2 will be considered case. Control women will be with BMI equals or less than 25 kg/m2.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2015-06; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
cardiac performance | 2 hours
  the cardiac performance (the left ventricular functions) in obese and lean pregnant women throughout each trimester and six weeks postpartum.

SECONDARY OUTCOMES:
The prevalence of cardiac lesions. | 2 hours
  the presence of other unnoticed cardiac lesions among candidates
The need of any medications among obese pregnant women | 9 months
  if an echo cardiogram results necessitate prescribing medication for any obese pregnant woman
The need of any advanced investigation among obese pregnant women | 9 months
  if an echo cardiogram results necessitate initiating advanced investigation for any obese pregnant woman
The need of hospitalization among obese pregnant women | 9 months
  if an echo cardiogram results necessitate hospitalization for any obese pregnant woman
The need of termination of pregnancy among obese pregnant women | 9 months
  if an echo cardiogram results necessitate termination of pregnancy for any obese pregnant woman
Maternal pregnancy outcomes | 9 months
  weight gain, obstetric disorders type delivery, duration of childbirth, blood pressure evolution, postpartum complications

CONTACTS AND LOCATIONS:
Overall Officials: ahmed altraigey, Study Director — Benha University; haytham attya, Principal Investigator — Zagazig University; nuzhat amer, Principal Investigator — Armed Forces Hospitals, Southern Region, Saudi Arabia; Mohamed Kolkailah, Study Chair — Armed Forces Hospitals, Southern Region, Saudi Arabia; mohammed mesilhy, Principal Investigator — Armed Forces Hospitals, Southern Region, Saudi Arabia; mohammed attia, Principal Investigator — Armed Forces Hospitals, Southern Region, Saudi Arabia; mohammed shehri, Principal Investigator — Armed Forces Hospitals, Southern Region, Saudi Arabia
Locations (1):
- antenatal clinic of Armed Forces Hospital, Southern Region, Khamis Mushait, 'Asir Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No